CLINICAL TRIAL: NCT05021380
Title: Salivary Immune/Stress Biomarkers Among Children
Acronym: OPI2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: University Paris 7 - Denis Diderot (Other)
Responsible Party: Principal Investigator, Elzbieta Paszynska, Assoc. Prof., Poznan University of Medical Sciences
Other Study IDs: PUMS
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Stress, Emotional; Dental Anxiety; Dental Pain and Sensation Disorder; Cortisol; Hypersecretion
Keywords: saliva; biomarkers; cortisol; IgA; IgG; IgM; amylase; opiorphin
MeSH Terms: conditions — Stress, Psychological; Toothache; Sensation Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group: 50 generally healthy children diagnosed with dental pain as symptomatic irreversible pulpitis (SIP) or symptomatic apical periodontitis (SAP) aged from 6 to 12 years old will be included to the GROUP.
  Interventions: Other: GROUP

INTERVENTIONS:
Other: GROUP — Non-invasive diagnosis of dental pain, dental root canal treatment, salivary specimen collection from the first visit to next and the last during 4 weeks of dental care

SUMMARY:
Background: The use of easily accessible biomarkers for assessing young patients' health is important. This study's aim is a measuring stress/immune biomarkers in saliva of healthy school-age children and compare subgroups according to age, sex, stress perception in dental pain related to symptomatic irreversible pulpitis (SIP) and symptomatic apical periodontitis (SAP).

Material and methods: 50 children diagnosed with SIP and SAP aged from 6 to 12 years old will be treated with root canal treatment. Dental examination using DMF score and oral hygiene level will be performedby experienced dentists. Salivary samples will be collected three times: before treatment in day of first dental visit (1), after two weeks (2), and after next two weeks = 30 days (3). Additionally, pain and stress perception will be examined by VAS scale and questionnaires dedicated for children anxiety: Frankl behavior rating scale, Venham's anxiety and behavior rating scale. Salivary immunoglobullins A, G, M, opiorphin, free cortisol and amylase will be measured using commercially available ELISA kits. Results will assess which of the measured salivary biomarkers is related to stress and dental pain, suggesting its use for evaluating in non-invasive way in childhood.

DETAILED DESCRIPTION:
Psychological stress impairs homeostasis in many aspects, including immune dysregulation with important variability according to age and sex. Use of easily accessible biomarkers is of importance to assess these changes in fragile subjects, as for example children, especially in a context of exposure to childhood stress experience, when invasive sampling procedures may increase the psychic stress.

Saliva is a promising tool which has been used both for acute and chronic stress Several salivary immune biomarkers are now considered to be sensitive and reliable readouts of mental stress in adult patients, among them free cortisol, alpha-amylase (sAA) and secretory immunoglobulin IgA (sIgA), IgM, IgG and opiorphin (OPI).

These four biomarkers may be measured easily in saliva, but in variable amounts according to age and sex, as well as in response to psychological stress. The main objective of this exploratory study was therefore to compare salivary levels of opiorphin, cortisol, sAA, sIgA, IgM, IgG in two groups of healthy children, 6-12 years old, a developmental age critical to mental disorders and dental interventional treatment, with ELISA tests.

This study's aim is a measuring stress/immune biomarkers in saliva of healthy school-age children and compare subgroups according to age, sex, stress perception in dental pain related to symptomatic irreversible pulpitis (SIP) and symptomatic apical periodontitis (SAP).

Material and methods: 50 children diagnosed with SIP and SAP aged from 6 to 12 years old will be treated with root canal treatment. Dental examination using DMF score and oral hygiene level will be performedby experienced dentists. Salivary samples will be collected three times: before treatment in day of first dental visit (1), after two weeks (2), and after next two weeks = 30 days (3). Additionally, pain and stress perception will be examined by VAS scale and questionnaires dedicated for children anxiety: Frankl behavior rating scale, Venham's anxiety and behavior rating scale. Salivary immunoglobullins A, G, M, opiorphin, free cortisol and amylase will be measured using commercially available ELISA kits. Results will assess which of the measured salivary biomarkers is related to stress and dental pain, suggesting its use for evaluating in non-invasive way in childhood.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 6 - 12 y.o.
* complaint dental pain
* diagnosis of symptomatic irreversible pulpitis or symptomatic apical periodontitis
* assigned agreement to the informed consent form by parents/caregivers and children cooperation

Exclusion Criteria:

* use of analgesics or antibiotics prior 48 h before specimen collection
* having a systemic disease
* disorders interfering with salivary function or flow
* regular medication intake interfering with salivary function or flow
* having temporary infectious disease
* having neurodevelopmental dysfunction (e.g ADHD)
* lack of cooperation during dental visits
* inability to understand the content of the informed consent form by parents/caregivers and children

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be recruited at University dental clinic in Child and Adolescent Section, one experienced dentist will conduct all dental and salivary collection procedures.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
dental pain | 30 days
  Proportion of subjects showing no increase in dental pain
salivary biomarkers | 30 days
  Proportion of subjects showing no increase in salivary biomarkers
dental anxiety | 30 days
  Proportion of subjects showing no increase in stress perception

CONTACTS AND LOCATIONS:
Overall Officials: Elzbieta Paszynska, Prof, Principal Investigator — Poznan University of Medical Sciences, Poland; Yves Boucher, Prof, Study Chair — Université de Paris & Groupe Hospitalier Pitié Salpêtrière, 75006 Paris, France
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No
we do not plan any individual participant data available share to other researchers

REFERENCES:
- [Background] Paszynska E, Roszak M, Slopien A, Boucher Y, Dutkiewicz A, Tyszkiewicz-Nwafor M, Gawriolek M, Otulakowska-Skrzynska J, Rzatowski S, Dmitrzak-Weglarz M. Is there a link between stress and immune biomarkers and salivary opiorphin in patients with a restrictive-type of anorexia nervosa? World J Biol Psychiatry. 2020 Mar;21(3):220-229. doi: 10.1080/15622975.2019.1593502. Epub 2019 Apr 23. PMID 30880537
- [Background] Boucher Y, Braud A, Dufour E, Agbo-Godeau S, Baaroun V, Descroix V, Guinnepain MT, Ungeheuer MN, Ottone C, Rougeot C. Opiorphin levels in fluids of burning mouth syndrome patients: a case-control study. Clin Oral Investig. 2017 Sep;21(7):2157-2164. doi: 10.1007/s00784-016-1991-0. Epub 2016 Nov 10. PMID 27834029
- [Result] Slavish DC, Szabo YZ. The effect of acute stress on salivary markers of inflammation: a systematic review protocol. Syst Rev. 2019 May 2;8(1):108. doi: 10.1186/s13643-019-1026-4. PMID 31046830